CLINICAL TRIAL: NCT00511212
Title: Clinical Study of Intravenous Immunoglobulin (IVIG) in Combination Therapy With Antibacterial Agents for Surgical Site Infection of the Lower Digestive Tract
Brief Title: Intravenous Immunoglobulin in Combination Therapy With Antibacterial Agents for SSI of the Lower Digestive Tract
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No eligible patient.
Sponsor: Multicenter Clinical Study Group of Osaka, Colorectal Cancer Treatment Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCSGO-0701
Record Dates: First submitted 2007-08-01; First posted 2007-08-03 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2007-08

CONDITIONS: Peritonitis; Postoperative Complications
Keywords: severe peritonitis; SSI; lower digestive tract surgery; Severe peritonitis after lower digestive tract surgery
MeSH Terms: conditions — Peritonitis; Postoperative Complications | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: intravenous immunoglobulin

SUMMARY:
The purpose of this study is to assess the clinical usefulness of IVIG in combination therapy with antibacterial agents for severe peritonitis after lower digestive tract surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients who have obvious symptoms and observation of post-surgical peritonitis, and meet the criteria described bellow.

1. Patients with >=38 degrees C, >=15,000/mm3 or <=3,000/mm3 of WBC and >=10mg/dL of CRP
2. Patients who have no abscess on the abdominal image
3. Patients who were administered antibacterial agents for 1 day or more, and show no sign of improvement
4. Patients who are 20 years old or older
5. Patients who have signed the agreement for participation in this study

Exclusion Criteria:

1. Patients who have a history of hypersensitivity to any of the ingredients of Immunoglobulin products
2. Patients who have a history of shock due to any of the ingredients of Immunoglobulin products
3. Patients who were administered immunoglobulin within 1 month before entry
4. Patients who were administered antibacterial agents for 1 day or more, and show signs of improvement
5. Patients with IgA deficiency
6. Patients with hereditary fructose intolerance
7. Patients with history of allergy or adverse effect for antibacterial agents
8. Patients who have underlying or concomitant disease that may seriously affect the assessment of this study
9. Patients who are or could be pregnant
10. Patients who have noninfectious fever, fungal infection or viral illness
11. Other patients who are judged to be inadequate to participate in this study by their physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-08; Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
clinical efficacy | at day 7

SECONDARY OUTCOMES:
clinical efficacy, recurrence rate, mortality, time between drug administration and defervescence, defervescence rate,time between drug administration and disappearance of clinical symptoms, improvement rate on clinical symptoms | at day 3 and at the end of test drug administration,

CONTACTS AND LOCATIONS:
Overall Officials: Morito Monden, MD, PhD, Study Chair — Multicenter Clinical Study Group of Osaka
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan